CLINICAL TRIAL: NCT04452825
Title: Cancer and Aging Reflections for Elders (CARE): A Geriatric-Specific Psychotherapy for Older Adults With Cancer
Brief Title: A New Psychotherapy Intervention for Older Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-191
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: geriatric cancer; geriatric specific; older adults with cancer; Psychotherapy; Memorial Sloan Kettering Cancer Center; 20-191
MeSH Terms: conditions — Neoplasms | interventions — elderberry extract; Methods; Social Work

STUDY DESIGN:
Intervention Model Description: This study is designed to test CARE delivered by telephone to improve cancer care for the population of older adults in a larger two-arm Randomized Controlled Trial (RCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer and Aging: Reflections for Elders (CARE) Intervention (Experimental): Session content and timing was developed and confirmed in our qualitative work (Expert Panel) and the CARE pilot study. Five sessions (45-60 minutes each) will be delivered over an 8-week period (+4 weeks). Following these sessions, four brief booster sessions (20-30 minutes each) will be delivered at a rate of approximately one per month to extend the interventions to 6 months (+3 months).
  Interventions: Behavioral: Cancer and Aging: Reflections for Elders (CARE) Intervention
- Social Work and Supportive Counseling (SWSC) (Experimental): The SWSC will include a social work assessment and follow-up augmented with additional components of supportive psychotherapy that have been shown to be an effective form of treatment for patients with cancer. Five sessions (45-60 minutes each) will be delivered over an 8-week period (+4 weeks). Following these sessions, four brief booster sessions (20-30 minutes each) will be delivered at a rate of approximately one per month to extend the interventions to 6 months (+3 months).
  Interventions: Behavioral: Social Work and Supportive Counseling (SWSC) Intervention

INTERVENTIONS:
Behavioral: Cancer and Aging: Reflections for Elders (CARE) Intervention — For full participants (not training case participants) five sessions (45-60 minutes each) will be delivered over an 8-week period (+4 weeks). Following these sessions, four brief booster sessions (20-30 minutes each) will be delivered at a rate of approximately one per month to extend the interventions to 6 months (+3 months).
  Arms: Cancer and Aging: Reflections for Elders (CARE) Intervention
Behavioral: Social Work and Supportive Counseling (SWSC) Intervention — The SWSC will include a social work assessment and follow-up augmented with additional components of supportive psychotherapy that have been shown to be an effective form of treatment for patients with cancer. For full participants (not training case participants) five sessions (45-60 minutes each) will be delivered over an 8-week period (+4 weeks). Following these sessions, four brief booster sessions (20-30 minutes each) will be delivered at a rate of approximately one per month to extend the interventions to 6 months (+3 months). Training case participants will follow a slightly condensed schedule.
  Arms: Social Work and Supportive Counseling (SWSC)

SUMMARY:
This study is being done to see if a new psychotherapy intervention called Cancer and Aging: Reflections for Elders (CARE) can effectively treat depression and distress in older cancer patients. CARE is a 5-session intervention that takes place over the phone. This study will compare CARE with the Social Work and Supportive Counseling (SWSC) intervention, which also takes place over the phone. SWSC is a standard psychotherapeutic intervention that has been shown to be a supportive and effective form of treatment for distress for patients with cancer. The researchers will look at which intervention is more effective in treating depression and distress in participants.

ELIGIBILITY:
Inclusion Criteria:

* As per self-report or medical record, ≥ 70 years of age
* As per self-report or medical record, has a diagnosis of cancer
* As per self-report or medical record, receiving active treatment (e.g., radiation, chemotherapy, hormone); OR received active treatment in the past 6 months (N/A for training case participants); OR are currently on active surveillance with follow-ups at least approximately every 6 months
* Received a HADS-D score of ≥ 6 or HADS-A score of ≥ 6 or a score of ≥ 4 on the distress thermometer. (N/A for training case participants)
* Received a Karnofsky Performance Rating Scale (KPRS) score of ≥ 60 (N/A for training case participants)
* Received a Blessed Orientation-Memory-Concentration Scale (BOMC) score of ≤ 11 (N/A for training case participants)
* Fluent in English, as per self-reported fluency of "well" or "very well"*

Exclusion Criteria:

* As per self-report, currently taking antidepressant medication for < 3 months
* As per self-report, currently receiving hospice care
* In the judgment of the consenting professional is unable to provide informed consent and complete study sessions and assessment
* As per self-report or as documented in the medical record, current untreated (e.g., no medication, no therapy) major psychotic disorder (schizotypal personality disorder, schizophreniform disorder, schizoaffective disorder). Patients diagnosed with a major psychiatric disorder will be reviewed by the study PI to determine eligibility prior to consent.

  * Language verification: Prior to enrollment, patients will be asked the following two questions by research staff to verify English fluency necessary for participation in the study:

    1. How well do you speak English? (must respond "Well" or "Very well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
    2. What is your preferred language for healthcare? (must respond English)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 459 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Depression and Anxiety: Hospital Anxiety and Depression Scale (HADS) | 9 months
  This 14-item scale, which has been well tested in cancer populations including elderly patients with cancer, has depression and anxiety subscales of seven items each. It is considered particularly useful for patients with chronic disease because of the absence of somatic items that often confound the determination of psychiatric problems among the medically ill.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org